CLINICAL TRIAL: NCT02165930
Title: An Open Label, Single Dose, Randomized, Two Way Crossover Study to Estimate Oxycodone Relative Bioavailability in Healthy Volunteers Following Administration of PF 00345439 Formulation K 40 Mg Under Fasting Conditions With 40% Ethanol Compared With Water
Brief Title: Effects of Ethanol on Oxycodone Pharmacokinetics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Responsible Party: Sponsor
Organization: PainT (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B4501037
Record Dates: First submitted 2014-06-10; First posted 2014-06-18 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Bioavailability; oxycodone; ethanol interaction; healthy volunteers
MeSH Terms: interventions — Oxycodone; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental)
  Interventions: Drug: Oxycodone; Drug: Naltrexone
- Treatment B (Experimental)
  Interventions: Drug: Oxycodone; Drug: Naltrexone

INTERVENTIONS:
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation K, single dose, administered with water, under fasting conditions
  Arms: Treatment A
Drug: Naltrexone — Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before,and 12 hours after study drug administration).
  Arms: Treatment A
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation K, single dose, administered with 40% ethanol, under fasting conditions
  Arms: Treatment B
Drug: Naltrexone — Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Arms: Treatment B

SUMMARY:
To Estimate Bioavailability Of 40 Mg Doses Of Pf-00345439 Formulation K Under Fasting Conditions with 40% Ethanol Compared with Water in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* History of moderate alcohol consumption
* Total body weight exceeding 64 kg

Exclusion Criteria:

* Evidence or history of clinically significant disease.
* Positive urine drug test
* History of alcoholism or heavy alcohol consumption

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Concentration at time 24 hours (C24) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
Plasma Decay Half-Life (t1/2) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4501037&StudyName=Effects%20of%20Ethanol%20on%20Oxycodone%20Pharmacokinetics%20in%20Healthy%20Volunteers